CLINICAL TRIAL: NCT00975923
Title: Safe Critical Care: Testing Improvement Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Theodore Speroff, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VU050413; AHRQ U18 HS015934 (Other Grant/Funding Number: AHRQ U18 015934)
Record Dates: First submitted 2009-09-10; First posted 2009-09-14 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-12

CONDITIONS: Central Line-associated Bloodstream Infection (CLABSI); Ventilator Associated Pneumonia
Keywords: Quality Improvement; Critical Care; Collaboratives; Patient Safety; Tool Kit
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Quality Improvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collaborative Group (Experimental): Quality Improvement Virtual Learning Collaborative with Interactive Teleconferences and Tool Kit
  Interventions: Behavioral: Collaborative Group
- Tool Kit Group (Active Comparator): Tool Kit of Evidence-Based Guidelines, Education Seminars, and Aide for Quality Improvement Methods
  Interventions: Behavioral: Tool Kit

INTERVENTIONS:
Behavioral: Collaborative Group — In addition to the Tool Kit materials and web site support, facility leaders and managers in this group agreed to participate in a Collaborative to improve critical care. The Collaborative differed from the IHI BTS model in that teams did not come together for face-to-face educational and planning sessions but instead attended web seminars and teleconferences. Between these "virtual" learning sessions, teams implemented some of the suggested change ideas, measured the results of those changes, and reported back to the larger group. Teams were supported through monthly educational and troubleshooting conference calls, individual coaching by faculty members, and an e-mail listserver designed to stimulate interaction among teams.
  Other Names: Collaborative Breakthrough Groups; Collaborative Quality Improvement Groups
  Arms: Collaborative Group
Behavioral: Tool Kit — Hospitals received a tool kit:evidence-based guidelines, CLABSI/VAP fact sheets, change ideas,quality improvement and teamwork methods, standardized data collection and charting tools. Periodic reminders of their commitment to the Safe Critical Care Initiative and access to web site containing all of the educational seminars, clinical tools, and quality improvement tools. ICUs in this group were on their own to initiate and implement a local hospital quality improvement initiative preventing CLABSI and VAP.
  Other Names: Quality Improvement
  Arms: Tool Kit Group

SUMMARY:
One group of hospitals participated in a collaborative approach for healthcare quality improvement while another group was provided only a tool kit. The investigators' objective was to determine if the Collaborative would perform better at preventing central line-associated bloodstream infections (CLABSI) and ventilator-associated pneumonias (VAP). Hospitals were randomized to the Tool Kit or Collaborative conditions. The investigators' study evaluated the effects on care processes and outcomes of a multi-institutional quality improvement initiative focused on preventing hospital associate infections. The investigators' hypothesis was that the strategies for implementing safe critical care practice will differ in level of achievement whereby the Collaborative group will perform better than the Tool Kit group. The outcome measure comprised clinical event rates and an index of safe practices that represent a bundling of key process measures related to evidence-based practices for preventing catheter-related blood-stream infections and ventilator-associated pneumonia in the intensive care unit.

DETAILED DESCRIPTION:
Continuous quality improvement (CQI) methodologies provide a framework for initiating and sustaining improvements in complex systems.1 By definition, CQI engages frontline staff in iterative problem solving using plan-do-study-act cycles of learning, with decision-making based on real-time process measurements. The Institute for Healthcare Improvement (IHI) has sponsored Breakthrough Series (BTS) Collaboratives since 1996 to accelerate the uptake and impact of quality improvement. These collaboratives are typically guided by evidence-based clinical practice guidelines, incorporate change methodologies, and rely on clinical and process improvement subject matter experts. Organizations have been adopting the collaborative model, and there is a growing literature on its positive impact. This collaborative approach to healthcare improvement has appealing face validity but lacks definitive evidence of its effectiveness. A recent derivative of collaboratives has been deployment of tool kits for quality improvement. Intuition suggests that such tools kits may help to enable change, and, thus some agencies advocate the simpler approach of disseminating tool kits as a change strategy. We sought to compare the collaborative model with the tool kit model for improving care. Recommendations and guidelines for central line-associated bloodstream infection (CLABSI) and ventilator-associated pneumonia (VAP) prevention have not been implemented reliably, resulting in unnecessary ICU morbidity and mortality and fostering a national call for improvement. Our study evaluated the effects on care processes and outcomes of a multi-institutional quality improvement initiative focused on preventing CLABSI and VAP in the intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* Medical centers with at least one adult or pediatric ICU.
* Medical centers within the Hospital Corporation of America (HCA) were eligible for enrollment.

Exclusion Criteria:

* Nonresponse to invitation to participate in our Safe Critical Care Initiative.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Speroff, PhD, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- HCA Hospital Corporation of America, Nashville, Tennessee, United States

REFERENCES:
- [Result] Talbot TR, Tejedor SC, Greevy RA, Burgess H, Williams MV, Deshpande JK, McFadden P, Weinger MB, Englebright J, Dittus RS, Speroff T. Survey of infection control programs in a large national healthcare system. Infect Control Hosp Epidemiol. 2007 Dec;28(12):1401-3. doi: 10.1086/523867. Epub 2007 Nov 1. PMID 17994522
- [Result] Wall RJ, Ely EW, Talbot TR, Weinger MB, Williams MV, Reischel J, Burgess LH, Englebright J, Dittus RS, Speroff T, Deshpande JK. Evidence-based algorithms for diagnosing and treating ventilator-associated pneumonia. J Hosp Med. 2008 Sep;3(5):409-22. doi: 10.1002/jhm.317. PMID 18951395
- [Result] Patel RP, Gambrell M, Speroff T, Scott TA, Pun BT, Okahashi J, Strength C, Pandharipande P, Girard TD, Burgess H, Dittus RS, Bernard GR, Ely EW. Delirium and sedation in the intensive care unit: survey of behaviors and attitudes of 1384 healthcare professionals. Crit Care Med. 2009 Mar;37(3):825-32. doi: 10.1097/CCM.0b013e31819b8608. PMID 19237884
- [Result] France DJ, Greevy RA Jr, Liu X, Burgess H, Dittus RS, Weinger MB, Speroff T. Measuring and comparing safety climate in intensive care units. Med Care. 2010 Mar;48(3):279-84. doi: 10.1097/MLR.0b013e3181c162d6. PMID 20125046
- [Result] Speroff T, Ely EW, Greevy R, Weinger MB, Talbot TR, Wall RJ, Deshpande JK, France DJ, Nwosu S, Burgess H, Englebright J, Williams MV, Dittus RS. Quality improvement projects targeting health care-associated infections: comparing Virtual Collaborative and Toolkit approaches. J Hosp Med. 2011 May;6(5):271-8. doi: 10.1002/jhm.873. Epub 2011 Feb 10. PMID 21312329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Leaders of all medical centers with at least 1 adult or pediatric ICU received an invitation to participate in a Quality Improvement initiative. Hospitals willing to participate were matched on geographic location and ICU volume and then randomized into either the Collaborative or Tool Kit Group in December 2005.
Groups:
- Collaborative Group: One group of hospitals is randomly allocated to the Collaborative Group
- Tool Kit Group: One group of hospitals is allocated randomly to the Tool Kit Group
Period: Overall Study
Arm/Group | Collaborative Group | Tool Kit Group
Started | 30 | 30
Completed | 30 | 29 (1 hospital was sold, yielding 29 hospitals in the Tool Kit Group)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Unit of analysis is Hospital and ICU
Groups:
- Total: Total of all reporting groups
Arm/Group | Collaborative Group | Tool Kit Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Number; unit: Hospitals] — Participants reporting whether ICU is pediatric (Age < 18 years) or adult (Age > 18 years) on baseline survey
  Hospitals
    Pediatric ICU (Age < 18 years) | 0 | 0 | 0
    Adult ICU (Age >= 18 years) | 30 | 30 | 60
Sex/Gender, Customized [Mean (Standard Deviation); unit: Percentage of ICU female patient volume] — baseline survey, percent of ICU patient volume that is female
  Percentage of ICU female patient volume
    Average % Female | 49.7 (5.7) | 50.3 (7.7) | 50 (6)
ICU annual patient volume [Median (Inter-Quartile Range); unit: ICU patients/year] — Patient volume was collected by a baseline survey of each participating hospital
  ICU patients/year | 568 [294 to 904] | 578 [244 to 1077] | 570 [250 to 950]
ICU mortality rate [Mean (Standard Deviation); unit: ICU mortality rate/year] — Annual ICU mortality rate provided by baseline survey among participating hospitals
  ICU mortality rate/year | 5.7 (3.1) | 7.1 (3.6) | 6 (3.5)
Medicare case-mix weight [Mean (Standard Deviation); unit: Medicare Case-Mix Index/year] — Average Medicare Case-Mix Index for annual ICU patient volume collected by baseline survey of participating hospitals. Patients are assigned to Medicare Severity-Diagnosis Related Groups (MS-DRG) based on principal and secondary diagnoses, age, procedures performed, co-morbidity, complications, discharge status, and gender. Each MS-DRG has a numeric weight that indicates the amount of resources required to treat patients in the group. The index, the average of the MS-DRG weights, measures the relative cost needed to treat the case-mix of patients in a hospital during the calendar year.
  Medicare Case-Mix Index/year | 1221 (1007) | 1295 (1110) | 1250 (1000)

OUTCOME MEASURES:

1. Primary Outcome: CLABSI and VAP Rates
Description: Central line associated bloodstream infections(CLABSI) and ventilator associated pneumonias (VAP) using Centers for Disease Control and Prevention definitions as number of events per 1,000 device days, data collection and surveillance methods.
Time Frame: 18 Months: 3-month baseline and quarterly post-intervention periods
Population: A cluster randomized trial randomly assigned hospitals to either the Collaborative or Tool Kit groups, stratified by region within the United States and ICU volume. Implementation and analysis was at the level of the ICU. One of the 30 hospital in the Tool Kit Group was sold, leaving 29 hospitals. Analysis was conducted per protocol.
Measure: Median (Inter-Quartile Range); unit: events/1000 device days
Groups:
- Collaborative Group: Hospitals randomly allocated to the Virtual Collaborative involving teleconferences and Tool Kit
- Tool Kit Group: Hospitals allocated randomly to the Tool Kit containing evidence-based guidelines and aides for conducting quality improvement
Arm/Group | Collaborative Group | Tool Kit Group
Number analyzed (Participants) | 30 | 29
events/1000 device days
  Baseline CLABSI | 1.84 [0 to 3.83] | 2.42 [0.65 to 6.80]
  3 Month CLABSI | 2.24 [0.54 to 4.69] | 2.47 [1.48 to 5.35]
  6 Month CLABSI | 2.28 [0.0 to 3.73] | 2.54 [0.0 to 4.98]
  12 month CLABSI | 1.18 [0.0 to 2.71] | 1.17 [0.0 to 3.61]
  18 Month CLABSI | 2.76 [0.0 to 4.67] | 1.16 [0.0 to 5.46]
  Baseline VAP | 2.14 [0.0 to 6.09] | 3.49 [0.0 to 7.04]
  3 Month VAP | 3.01 [0.0 to 9.11] | 3.32 [0.0 to 8.25]
  6 Month VAP | 2.72 [0.0 to 7.09] | 4.61 [0.0 to 9.37]
  12 Month VAP | 2.67 [0.0 to 4.47] | 2.66 [0.0 to 4.82]
  18 Month VAP | 2.93 [0.0 to 7.63] | 2.06 [0.0 to 6.59]
Statistical Analysis 1: Comparison: Collaborative Group vs Tool Kit Group; Infection rates were analyzed using hierarchical negative binomial regression models to model infection rate changes over time and account for clustering of ICUs within hospitals and adjusting for baseline covariates. Power was calculated a priori with a 1-tailed alpha of 0.05 and group size of 30; a 50% decrease in infection rates in the Collaborative group and 15% for the Tool Kit group, yielding power ranging from 82% to 91% for testing group differences; Test type: Superiority or Other; p < .05, Regression, Linear — p-value and confidence intervals; infection rates per device days = 2.00, 95% CI 2-sided [1.0 to 3.0], Standard Error of Mean .05

2. Secondary Outcome: Access of Tools and Use of Quality Improvement Strategies
Description: Follow-up survey of ICU nurse and quality managers for all participating medical centers from Jan 2008 through April 2008 included questions about the implementation of process interventions: Access and use of clinical guidelines tools, access and use of quality improvement tools, and types of quality improvement implementation strategies.
Time Frame: 18 months
Population: per protocol
Measure: Number; unit: Percentage of ICUs
Groups:
- Tool Kit Group: Hospitals allocated randomly to only a Tool Kit of clinical guidelines and aides for quality improvement
Arm/Group | Collaborative Group | Tool Kit Group
Number analyzed (Participants) | 26 | 19
Percentage of ICUs
  Clinical Tool Use | 61 | 49
  Data Tools | 56 | 30
  Strategies | 69 | 54
Statistical Analysis 1: Comparison: Collaborative Group vs Tool Kit Group; It was hypothesized that the Collaborative group would engage in more processes and tools than the Tool Kit group. Power was based on infection rates; Test type: Superiority or Other; p < 05, Chi-squared; percentages = 10 — Power calculation used alpha = .05 and group size = 30.The estimated effect was a 50% decrease in infection rates for the Collaborative Group and from 10% to 15% decrease in the Tool Kit group.Power ranged from 82%-91% for testing group differences

ADVERSE EVENTS:
Time Frame: No other adverse event data were collected other than the primary study outcomes
Description: 0 hospital (ICU) participants were at risk as no other adverse events were collected or assessed other than the primary study outcomes.
Groups:
- Collaborative Group: Hospitals allocated randomly to the Collaborative Quality Improvement intervention with teleconferences and Tool Kit
- Tool Kit Group: Hospitals allocated randomly to the Tool Kit containing evidence-based guidelines and aides for quality improvement
Arm/Group | Collaborative Group | Tool Kit Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29

LIMITATIONS AND CAVEATS:
Each participant tailored their interventions; we were not able to test the components of CQI. Data were dependent on self-reports. Our collaborative was virtual and does not address benefits from face-to-face networking of large scale projects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No